CLINICAL TRIAL: NCT03574935
Title: Clinical Evaluation and Generalized Application of "Qing-Hua-Bu" Three Dynamic Sequential Therapy of Diabetic Ulcer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16411955000
Record Dates: First submitted 2018-06-09; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Diabetic Foot; Ulcer, Skin
Keywords: "Qing-Hua-Bu"; Dynamic sequential treatment; Clinical evaluation; Generalized application
MeSH Terms: conditions — Diabetic Foot; Skin Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Chinese medicine (Experimental): External Chinese medicine include 3 kinds of formula，including:
  Qin, Hua and Bu will be applied to cover the participants' lesions in wet dressing form. Dosage form:5g/ml; frequency:qd; duration:2months.
  Interventions: Drug: External Chinese medicine; Drug: External Western medicine
- External Western medicine (Active Comparator): Ethacridine Lactate Solution, 1% Sulfadiazine Silver Cream and rb-bFGF will be applied to cover the participants' lesions. Dosage form:3g/ml; frequency:qd; duration: 2months.
  Interventions: Drug: External Chinese medicine; Drug: External Western medicine

INTERVENTIONS:
Drug: External Chinese medicine — External Chinese medicine:
  For patients in the treatment group, they will accept one of three specific External Chinese medicine according to their lesions and corresponding syndromes:
  1. Chinese herb of "Clear heat-Remove dampness-Detoxicate" for patients belong to heat syndrome;
  2. Chinese herb of "Activating blood-Removing stasis" for patients belong to stasis syndrome;
  3. Chinese herb of "Supplement deficiency-Generate muscles" for patients belong to deficiency syndrome.
  Other Names: "Qing-Hua-Bu" Three Dynamic Sequential Therapy
Drug: External Western medicine — For patients in the control group, they will accept one of three specific external Western medicine according to their lesions:
  1.Ethacridine Lactate Solution(lesions with much effusion)； 2.1% Sulfadiazine Silver Cream（lesions with infection）； 3.rb-bFGF(lesions with no slough and look clear).
  Other Names: No.

SUMMARY:
This project is based on investigator team's ten year experience on diabetic ulcer and goes on further developing basic research and concluding clinical experience. The investigator team has recently developed "Remove stasis to generate granulation tissue" into "Remove slough to generate granulation tissue". Investigators have applied the principle of "Remove stasis" in the medium and later stage of treatment to make "Remove slough-Eliminate stasis-Generate granulation tissue" become the basic principle of three-stage sequential treatment. Investigators will further conclude Chinese medicine therapy in the stage of "Qing-Hua-Bu" and evaluate safety, applicability and availability of it. Therefore, the research can help improve clinical diagnosis and treatment technique and transfer the study result of Chinese medicine experience on diabetic ulcer.

DETAILED DESCRIPTION:
Aim: Under guidance of "Clear pus-Remove stasis-Supplement muscles" theory, to observe clinical effectiveness of dynamic Chinese external therapy of "Qing-Hua-Bu" in treating diabetic ulcer and partially explain potential wound healing mechanism.

Method: Clinical observation: To adopt the design method of open and parallel control test and include 150 diabetic ulcer patients. The treatment group was supplied with external clearing heat, removing stasis and supplementing deficiency Chinese medicine, while the control group was supplied with sulfadiazine silver cream, furacilin solution and bovine basic fibroblast growth factors (b-FGF) spray. To perform the dressing change for wound every day and persist in dressing change for two months. To record dynamic wound healing progress by digital camera. After finishing course, to compare wound healing, pus, exudate, granulation tissues and epithelial tissues and analyze these data by SPSS22.0.

ELIGIBILITY:
Inclusion Criteria:

1. accord with standard of syndrome differentiation of traditional Chinese medicine and western medicine diagnostic criteria;
2. age between 18-65 years old, gender, ethnic unlimited;
3. agreed to participate in clinical trials can observe and cooperate with the visitor on schedule;
4. sign the informed consent form and mark the date;
5. If the patients are in the child-bearing period, they should accept the test of HCG and the result should be negative;

Exclusion Criteria:

1. systematic application of steroids or immunosuppressor within 2 weeks;
2. be allergic to any contents of known studied medicine;
3. experiment results that may influence patients' safety;
4. women within gestation period，suckling period or planning to gestation period;
5. patients with severe heart, liver or kidney diseases;
6. have received other studying medicine or taken part in other clinical experiments;
7. cannot cooperate with the study for any reasons,such as language understanding and not able to see the doctors;
8. other situations or diseases that researchers think may bring obvious risks to patients or interfere with the study results.
9. cancer ulcer; tuberculotic ulcer；radioactive ulcer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing rate | up to 56 days after treatment
  To perform the dressing change for wound every day and persist in dressing change for two months. To record dynamic wound healing progress by digital camera. After finishing course, to compare wound healing, pus, exudate, granulation tissues and epithelial tissues and analyze these data by SPSS22.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Study Chair — Department of dermatology, Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai